CLINICAL TRIAL: NCT04475562
Title: Can the Electronic Nose Smell COVID-19? A Proof-of-principle Study
Brief Title: Can the Electronic Nose Smell COVID-19?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Nicole Bouvy, Prof. Dr. Nicole D. Bouvy, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: eNoseCOVID
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: Electronic nose; Volatile organic compounds; Diagnosis
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 suspected (Other): Participants were recruited at the outpatient clinic for MUMC+ employees with COVID-19 symptoms or at the nursing unit where a SARS-CoV-2 patient was admitted.
  Interventions: Device: Aeonose

INTERVENTIONS:
Device: Aeonose — All participants breathed through the Aeonose for five minutes. This device contains metal-oxide sensors that change in conductivity upon reaction with VOCs in exhaled breath. These conductivity changes are input data for machine-learning and used for pattern recognition. A nose clip was placed on the nose of each participant to avoid entry of non-filtered air in the device. Before measuring, the Aeonose was flushed with room air, guided through a carbon filter as well. During each measurement, a video was displayed to distract the participant and to reduce the chance of hyperventilation. Failed breath tests were excluded from analysis; the reason for failure was documented. Four similar Aeonose devices were used for breath analysis. A full-measurement procedure required sixteen minutes.

SUMMARY:
Infection with SARS-CoV-2 causes Corona Virus Disease (COVID-19). The most standard diagnostic method is reverse transcription-polymerase chain reaction (RT-PCR) on a nasopharyngeal and/or an oropharyngeal swab. The high occurrence of false-negative results due to the non-presence of SARS-CoV-2 in the oropharyngeal environment renders this sampling method not ideal. Therefore, a new sampling device is desirable. This proof-of-principle study investigates the possibility to train machine-learning classifiers with an electronic nose (Aeonose) to differentiate between COVID-19 positive- and negative persons based on volatile organic compounds (VOCs) analysis.

Methods: between April and June 2020, participants were invited for breath analysis when a swab for RT-PCR was collected. If the RT-PCR resulted negative, presence of SARS-CoV-2 specific antibodies was checked to confirm the negative result. All participants breathed through the Aeonose for five minutes. This device contains metal-oxide sensors that change in conductivity upon reaction with VOCs in exhaled breath. These conductivity changes are input data for machine-learning and used for pattern recognition. The result is a value between -1 and +1, indicating the infection probability.

ELIGIBILITY:
Inclusion Criteria:

* Participants of whom an oropharyngeal or nasopharyngeal swab was collected to perform RT-PCR on.

Exclusion Criteria:

* Participants who were experiencing dyspnea or needed supplemental oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
COVID 19 positive vs negative | 3 months
  Ability of the eNose to distinguish COVID-19 positive from COVID-19 negative persons based on VOC patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] de Lacy Costello B, Amann A, Al-Kateb H, Flynn C, Filipiak W, Khalid T, Osborne D, Ratcliffe NM. A review of the volatiles from the healthy human body. J Breath Res. 2014 Mar;8(1):014001. doi: 10.1088/1752-7155/8/1/014001. Epub 2014 Jan 13. PMID 24421258
- [Background] Schuermans VNE, Li Z, Jongen ACHM, Wu Z, Shi J, Ji J, Bouvy ND. Pilot Study: Detection of Gastric Cancer From Exhaled Air Analyzed With an Electronic Nose in Chinese Patients. Surg Innov. 2018 Oct;25(5):429-434. doi: 10.1177/1553350618781267. Epub 2018 Jun 18. PMID 29909757
- [Background] Bikov A, Lazar Z, Horvath I. Established methodological issues in electronic nose research: how far are we from using these instruments in clinical settings of breath analysis? J Breath Res. 2015 Jun 9;9(3):034001. doi: 10.1088/1752-7155/9/3/034001. PMID 26056127
- [Background] Bijland LR, Bomers MK, Smulders YM. Smelling the diagnosis: a review on the use of scent in diagnosing disease. Neth J Med. 2013 Jul-Aug;71(6):300-7. PMID 23956311
- [Background] van Geffen WH, Bruins M, Kerstjens HA. Diagnosing viral and bacterial respiratory infections in acute COPD exacerbations by an electronic nose: a pilot study. J Breath Res. 2016 Jun 16;10(3):036001. doi: 10.1088/1752-7155/10/3/036001. PMID 27310311